CLINICAL TRIAL: NCT02813252
Title: Long-Term Follow-up Protocol for Subjects Treated With JCAR015
Brief Title: Long-Term Follow-up Study for Patients Previously Treated With JCAR015
Status: Completed | Type: Observational
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: 015002
Record Dates: First submitted 2016-06-21; First posted 2016-06-24 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: long-term follow-up; chimeric antigen receptor (CAR) T cells; JCAR015
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA prepared from peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- JCAR015-treated: Patients who received previous treatment with JCAR015
  Interventions: Genetic: JCAR015

INTERVENTIONS:
Genetic: JCAR015 — No study drug is administered in this study. Patients who received JCAR015 in a previous trial will be evaluated in this trial for long-term safety and efficacy.

SUMMARY:
This study will provide long-term follow-up for patients who have received treatment with JCAR015 in a previous clinical trial. In this study, patients will be followed for up to 15 years after their last dose of JCAR015 for evaluation of delayed adverse events, presence of persisting JCAR015 vector sequences, and survival.

ELIGIBILITY:
Inclusion criteria:

* Patients who have received at least one dose of JCAR015 in a previous treatment protocol.
* Patients who have provided informed consent for the long-term follow-up study prior to study participation.

Exclusion criteria:

* None. All patients who have previously received JCAR015 treatment are eligible for this long-term follow-up study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously treated with JCAR015 in a prior clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with adverse events | Every year for up to 15 years post-treatment
Proportion of patients with detectable JCAR015 vector sequences during first 5 years post-treatment | Every 6 months for the first 5 years post-treatment
Proportion of patients with detectable JCAR015 vector sequences between 5 and 15 years post-treatment | Every year from 5 years post-treatment to up to 15 years post-treatment
Survival | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No